CLINICAL TRIAL: NCT05307549
Title: COVID-19 and Brain: Cognition and Mental Health
Acronym: DIANA
Status: Completed | Type: Observational
Sponsor: University of Barcelona (Other)
Collaborators: Consorci Sanitari de Terrassa (Other); Universitat Politècnica de Catalunya (Other)
Responsible Party: Principal Investigator, Carme Junqué, Professor, University of Barcelona
Other Study IDs: 2020PANDE00053
Record Dates: First submitted 2022-03-22; First posted 2022-04-01 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: COVID-19; Cognition; Mental Health; Neuroimaging; MachineLearning
MeSH Terms: conditions — COVID-19; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, Feces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-COVID patients: Adults survivors from severe COVID-19
- Controls: Healthy adult controls

SUMMARY:
The main goal of DIANA is to investigate the potential discriminative power of multimodal biomarkers in COVID adverse outcomes. The study of the neuropathological underlying mechanisms in COVID from a translational approach at: (1) the behavioural-clinical level from cognitive, emotional and functional data; (2) the brain connectome level from structural and functional imaging data; and (3) biogenetic level from blood and stool data. Moreover, the investigators will develop machine learning based predictive models of cognitive, mental health, functionality, and brain connectivity evolution in post-COVID syndrome patients.

DETAILED DESCRIPTION:
DIANA project is an observational, descriptive, and cross-sectional study in which participants will not be randomized. Case people (adult survivors of severe COVID-19 N=134) will compare to healthy adult controls (n=66). It is a multicentric study where all the participants will be recruited from eleven Catalan public health institutions. The participants will be assessed on cognitive, emotional and functional status. The investigators will obtain a blood sample to study inflammation, vascular risk, growth factors, angiogenesis, neurogenesis, and cellular metabolism biomarkers and genes, and a stool sample for gut microbiota study. Structural and functional MRI will be performed on a subgroup of participants 40 COVID-19 survivors and 40 healthy controls.

The objectives of the project are:

1. To examine the impact of the COVID-19 illness on cognition, emotion/behavior, and functionality.
2. To examine the possible affectation in brain grey and white matter and functional connectivity of severe forms COVID-19 survivors.
3. To relate demographic characteristics, previous pathologies, lifestyle, baseline cerebral status, genetic polymorphism, and clinical data in acute illness with cognitive, mental health, functionality, and brain connectivity outcomes of severe forms COVID-19 survivors.
4. To study the post-COVID-19 biomarkers of inflammation, vascular risk, growth factors, angiogenesis, neurogenesis, and cellular metabolism and its relationship with the cognitive, mental health, functionality, and brain connectivity outcomes of severe forms COVID-19 survivors.
5. To quantify the presence of different bacterial species in the post COVID stool sample and analyze the wealth and diversity of the diverse populations. To study if these values are related to the performance of neuropsychological and behavioral tests and neuroimaging data.
6. - To develop machine learning based predictive models of cognitive, mental health, functionality and brain connectivity evolution in post COVID 19 survivors.

ELIGIBILITY:
Post-COVID Group:

Inclusion Criteria:

* Confirmed diagnosis of COVID-19 according to WHO interim with signs and symptoms of the severe disease during the acute phase
* Presence of cognitive complaints after COVID-19 diagnosis
* Participants have to be discharged from the hospital at least three months before inclusion
* Accept to take part in the study and sign the informed consent according to the Declaration of Helsinki

Exclusion Criteria:

* Participants have symptoms of delirium according to Delirium Rating Scale-revised 98
* Established diagnosis before COVID-19 disease of psychiatric, neurological, neurodevelopmental disorder or systemic pathologies are known to cause cognitive deficits
* Motor or sensory alterations that impede the neuropsychological examination
* Participants with a metal prosthesis (for MRI studies)
* Subjects suffering from claustrophobia or requiring sedation due to high anxiety (for MRI studies)

Healthy Adult Control group

Inclusion Criteria

* Healthy people who have not had COVID-19
* Accept to take part in the study and sign the informed consent according to the Declaration of Helsinki

Exclusion criteria: the same as COVID-19 survivors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COVID-19 survivors group will be recruited in hospital and primary care services.
  The control population will be searched in the general population through primary care centers, the media, social networks, and they will be offered to participate in the study without remuneration.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Differences between groups in auditory attention | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Auditory attention is measured with Digit Span Forward. Participants are asked to repeat numbers in the same order as read aloud by the examiner. Higher scores mean a better outcome.
Differences between groups in working memory | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Working memory is measured with Digit Span Backward. Participants are asked to repeat the numbers in the reverse order of that presented by the examiner. Higher scores mean a better outcome.
Differences between groups in language | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Language is measured with the Boston Naming Test. It consists of 60 line drawings of objects of graded difficulty, ranging from very common things to less familiar objects. The total score is the sum of correct answers. Higher scores mean a better outcome.
Differences between groups in verbal memory | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Verbal memory is measured with the Auditory Verbal Learning Test (AVLT). It is a word-learning test where five presentations of a 15-word list are given, each followed by an attempted recall. This is followed by a second 15-word interference list (list B), followed by recall of list A. Delayed recall and recognition are also tested. Higher scores mean a better outcome.
Differences between groups in visual memory | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Visual memory is measured with the Rey-Osterrieth Complex Figure (ROCF) test. The participants are asked to copy complex geometric shapes and then reproduce them from memory. A delayed recall is also tested. Higher scores mean a better outcome.
Differences between groups in psychomotor speed | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Processing speed is measured with Coding subtest of WAIS. Participants are asked to use a key to put in the appropriate symbols for a list of numbers. Higher scores mean a better outcome.
Differences between groups in perceptual reasoning | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Perceptual reasoning is measured with Matrix reasoning subtest of WAIS. Participants are asked to choose which of some possible options the missing picture is from matrix of abstract pictures. Higher scores mean a better outcome.
Differences between groups in executive function | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  A composite score is made with the z-scores of phonemic (sum of the three letters) and semantic fluency, Trail Making Test B (time) and STROOP test (color-word interference total items in 120 seconds).
Differences between groups in social cognition | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Social cognition is measured with the Reading the Mind in the Eyes Test. Participants are asked to choose the emotional state that best describes the eyes, choosing between one of four possible emotions in the 36 photographs of male and female eyes depicting emotional states. Higher scores mean a better outcome.
Differences between groups in anxiety | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Anxiety is measured with the 7-item Generalized Anxiety Disorder Scale (GAD-7), a Likert-type scale with questions ranging from "not at all" (0 points) to "nearly every day" (3 points). The maximum score is 24. Higher scores mean a worse outcome.
Differences between groups in depression | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Depression is measured with the Patient Health Questionnaire-9 (PHQ-9) which scores each of the 9 DSM-IV criteria as "not at all" (0 points) to "nearly every day" (3 points). Higher scores mean a worse outcome.
Differences between groups in Post-traumatic Stress Disorder | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Post-Traumatic Stress Disorder is measured with The Post-Traumatic Stress Disorder Checklist (PCL-5), a 20-item questionnaire corresponding to the DSM-5 symptom criteria for PTSD, which scores each criterion as "not at all" (0 points) to "extremely" (4 points). The ratings of items are added together to calculate the total score (range=0-80). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Differences between groups in Fatigue | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Fatigue is measured with the Chalder Fatigue Scale, an 11-item questionnaire measuring the severity of physical and mental fatigue on two separate subscales. Seven items represent physical fatigue (items 1-7) and 4 represent mental fatigue (items 8-11). Each item " less than usual" (0) to " much more than usual" (3). The ratings of items are added together to calculate the total score (range=0-33). High scores represent high levels of fatigue.
Differences between groups in Quality of Life | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Quality of life is measured with a 12-item World Health Organization Disability Assessment Schedule-II (WHODAS-II). Patients are asked to state the level of difficulty experienced, considering how they usually do the activity. The scale scores each item as "none" (1) to "cannot do" (5). The total score is calculated with an SPSS syntax, and the range varies from 0 to 100, with higher scores reflecting more significant disability.
  (WHODAS-II)
Differences between groups in White Matter integrity | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  White matter integrity: tractography measured by MRI
Differences between groups in brain Volumetry | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Grey and white matter volume measured by MRI
Differences between groups in Resting-state connectivity | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Resting state brain activity using fMRI
Differences between groups in plasmatic Interleukin- 6 (IL-6) | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of IL-6 are measured with enzyme-linked immunosorbent assay (ELISA) Kit
Differences between groups in plasmatic D-Dimer | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of D-Dimer are measured with ELISA Kit
Differences between groups in plasmatic Nerve Growth Factor (NGF) | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of NGF are measured with ELISA Kit
Differences between groups in plasmatic Glial Fibrillary Acidic Protein (GFAp) | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of GFAp are measured with ELISA Kit
Differences between groups in plasmatic NT-proB-type Natriuretic Peptide (BNP) | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of BNP are measured with ELISA Kit
Differences between groups in plasmatic lipid peroxidation products | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of malondialdehyde are measured with TBARS assay method
Differences between groups in plasmatic Thrombomodulin | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of Thrombomodulin are measured with ELISA Kit
Differences between groups in plasmatic Endothelin 1 | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of Endothelin 1 are measured with ELISA Kit
Differences between groups in plasmatic Ferritin | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of Ferritin are measured with biochemical assay
Differences between groups in plasmatic C-Reactive Protein (CRP) | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of CRP are measured with high sensitivity c-reactive protein ELISA Kit
Differences between groups in Microbiota data | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Bacterial composition of stool samples in terms of relative abundance

CONTACTS AND LOCATIONS:
Overall Officials: Carme Junqué, PhD, Study Director — University of Barcelona
Locations (1):
- University of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carreras-Vidal L, Pacheco-Jaime L, Ariza M, Cano N, Garolera M, Garcia-Vicente C, Roura I, Capdevila-Lacasa C, Oltra J, Pardo J, Martin-Barcelo C, Campabadal A, Sala-Llonch R, Bargallo N, Barrue C, Bejar J, Cortes CU, Junque C; NAUTILUS-Project Collaborative Group; Segura B. Functional brain abnormalities in post COVID-19 condition and their relationship with cognition. Sci Rep. 2025 Jul 1;15(1):22259. doi: 10.1038/s41598-025-00739-3. PMID 40595626
- [Derived] Pacheco-Jaime L, Garcia-Vicente C, Ariza M, Cano N, Garolera M, Carreras-Vidal L, Roura I, Capdevila-Lacasa C, Oltra J, Pardo J, Martin-Barcelo C, Campabadal A, Sala-Llonch R, Bargallo N, Barrue C, Bejar J, Cortes CU, Junque C, Segura B; NAUTILUS-Project Collaborative Group. Structural brain changes in post-COVID condition and its relationship with cognitive impairment. Brain Commun. 2025 Feb 12;7(1):fcaf070. doi: 10.1093/braincomms/fcaf070. eCollection 2025. PMID 40008326
- [Derived] Ariza M, Cano N, Segura B, Adan A, Bargallo N, Caldu X, Campabadal A, Jurado MA, Mataro M, Pueyo R, Sala-Llonch R, Barrue C, Bejar J, Cortes CU; NAUTILUS Project Collaborative Group; Garolera M, Junque C. COVID-19 severity is related to poor executive function in people with post-COVID conditions. J Neurol. 2023 May;270(5):2392-2408. doi: 10.1007/s00415-023-11587-4. Epub 2023 Mar 20. PMID 36939932
- [Derived] Ariza M, Cano N, Segura B, Adan A, Bargallo N, Caldu X, Campabadal A, Jurado MA, Mataro M, Pueyo R, Sala-Llonch R, Barrue C, Bejar J, Cortes CU; NAUTILUS-Project Collaborative Group; Junque C, Garolera M. Neuropsychological impairment in post-COVID condition individuals with and without cognitive complaints. Front Aging Neurosci. 2022 Oct 20;14:1029842. doi: 10.3389/fnagi.2022.1029842. eCollection 2022. PMID 36337708